CLINICAL TRIAL: NCT06540677
Title: Use of Meludia to Evaluate the Benefits of Music Training in Cochlear Implant Users: a Randomized
Brief Title: Musical Training in Cochlear Implant Users
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Miryam Calvino, Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-5880
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Deafness; Perception, Bilateral
Keywords: Cochlear implant; Musical training; Auditory Perception; Speech Perception; Cognitive Function; Quality of life
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Musical training (MT Group) (Experimental): Based on the literature review, we will establish 20 minute sessions three times per week over a period of 4 weeks for participants in the MT group. After this period, all the participants will be evaluated (session 1). An additional training period of 12 weeks, also with 20-min sessions three times per week, will then be conducted in the MT group, followed by another evaluation (session 2).
  In sessions 0 (at enrollement), 1, and 2, they will complete the MuRQoL or MuQPP to evaluate their exposure to music and the AQoL-8D to evaluate their quality of life. Further, they will perform the "Listen up" test, the cognition tests, and the audiological tests in quiet and in noise.
  Interventions: Other: Musical training
- Non Musical training (NMT Group) (No Intervention): Participants won't perform musical training. In sessions 0 (at enrolment), after 4 weeks , and again after 12 additional weeks, they will complete the MuRQoL or MuQPP to evaluate their exposure to music and the AQoL-8D to evaluate their quality of life. Further, they will perform the "Listen up" test, the cognition tests, and the audiological tests in quiet and in noise.

INTERVENTIONS:
Other: Musical training — Musical training with Meludia software, an online self-paced music training application
  Arms: Musical training (MT Group)

SUMMARY:
With this protocol we want to investigate the degree to which the use of Meludia training (the online self-paced music training application) can improve music perception, music enjoyment, and speech understanding in pediatric and postlingually deafened adult CI users. The study also aims to assess the participants' changes in cognitive skills (attention and memory) and quality of life.

Participant recruitment Group A: New CI users All postlingually deafened patients older than 6 years who undergo cochlear implantation at the La Paz Hospital in Madrid (Spain) between September 2024 and September 2027 will be invited to participate in the study.

Group B: Experienced CI users CI users older than 6 years old with at least 12 months of stable fitting will be recruited from the CI program at the La Paz Hospital between September 2024 and September 2027. Within this group this group, it will be required that pediatric CI have been implanted before the age of 3 years.

Both in the Group A and in the Group B, participants at the time of enrolment will be randomly divided 1:1 into two groups, with subjects being instructed to practice with Meludia music training application (intervention group: MT group) and participants in the non-MT group non receiving music training (NMT group).

We will establish 20 minute sessions three times per week over a period of 4 weeks for participants in the MT group. After this period, all the participants will be evaluated (session 1). An additional training period of 12 weeks, also with 20-min sessions three times per week, will then be conducted in the MT group, followed by another evaluation (session 2).

The ongoing protocol for music training cannot replace conventional tools in the rehabilitation of CI users. However, after scientific-based improvement of music practice protocols (easily implementable, low-priced, and with little probability of adverse effects) as an auditory practice rehabilitation along with the conventional methods, music training may provide an important tool for the aural rehabilitation plan

ELIGIBILITY:
Inclusion Criteria:

* Group A: New CI users All postlingually deafened patients older than 6 years who undergo cochlear implantation at the La Paz Hospital in Madrid (Spain) between September 2024 and September 2027 will be invited to participate in the study.

Group B: Experienced CI users CI users older than 6 years old with at least 12 months of stable fitting will be recruited from the CI program at the La Paz Hospital between September 2024 and September 2027. Within this group this group, it will be required that pediatric CI have been implanted before the age of 3 years.

All participants in both groups will have been implanted either unilaterally or bilaterally with CI devices from the manufacturer MED-EL (Innsbruck, Austria).

Exclusion Criteria:

* Participants will be excluded from the study if they have visual or motor impairments that prevent them from seeing the computer screen and pressing the correct keys, or if there is evidence of cognitive decline. Participants who have previously used Meludia software will also be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Score obtained to evaluate the effects of music training in music perception | 12 weeks
  "Listen Up" music exercises will be used to evaluate music perception
Score obtained to evaluate the effects of music training in music enjoyment | 12 weeks
  1. MuRQoL (Music Related Quality of Life) questionnaire will be used to quantify both the frequency and importance of music in adults CI users. Score: 0-5, higher results means better performance
  2. The Music Questionnaire for Pediatric Population will be used to quantify music enjoyment in children with CI. Score: 0-10, higher results means better performance

SECONDARY OUTCOMES:
Score obtained to evaluate the effects of music training in speech perception | 12 weeks
  1. Disyllables in silence will be used to evaluate speech perception in CI users (0-100%).
  2. Matrix test will be used to evaluate speech perception in noise in adults with CI.
  Higher results means better performance
Score obtained to evaluate the effects of music training in cognitive skills | 12 weeks
  1. Mini Mental State Examination will be used to assess cognitive skills in adult CI users.
  2. The Performance intelligence quotient and the Wechsler intelligence scale for children will be used to assess cognitive skills in children with CI Higher results means worse cognitive skills
Score obtained to evaluate the effects of music training in quality of life | 12 weeks
  1.The AQoL-8D (Assessment of Quality of Life-8 dimentions) questionnaire will be used to assess. individual's quality of life in adult CI users.
  Score: 1.00 (full health) to 0.00 (death-equivalent health states) to -0.04 (health states worse than death)

CONTACTS AND LOCATIONS:
Overall Officials: Miryam Calvino, Principal Investigator — La Paz University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvino M, Gavilan J, Lassaletta L. Use of Meludia to evaluate the effect of music training in cochlear implant users: study protocol of a randomised controlled study. BMJ Open. 2025 Apr 25;15(4):e092207. doi: 10.1136/bmjopen-2024-092207. PMID 40280615